CLINICAL TRIAL: NCT03714958
Title: A Single-center, Phase 1 Dose Escalation Study of Trametinib Combined With HDM201 in Patients With RAS/RAF Mutant and TP53 Wild-type Advanced/Metastatic Colorectal Cancer.
Brief Title: Trametinib + HDM201 in CRC Patients With RAS/RAF Mutant and TP53 Wild-type Advanced/Metastatic Colorectal Cancer Mutant and TP53 Wild-type
Acronym: TRAHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET17-063 (TRAHD)
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — siremadlin; trametinib

STUDY DESIGN:
Intervention Model Description: This study will utilize sequential and adaptive Bayesian design using the method of Time-to-event Continual Reassessment Method (CRM) to guide dose escalation and estimate the MTD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination HDM201 - Trametinib (Experimental): * HDM201: Therapeutic class HDM2 inhibitor, given Per Os every D1 and D8 over a 28 day cycle. Four dose-levels possible in dose escalation part: 40 mg, 80mg, 100 mg, 120mg.
  * Trametinib: Therapeutic class Protein kinase inhibitor of MEK1 and MEK2 activation and kinase activity. Administrated daily, countinous dosing , twodose-level possible in dose escalation: 1.5 mg and 2mg
  Interventions: Drug: HDM201; Drug: Trametinib

INTERVENTIONS:
Drug: HDM201 — Treatment will be administered as long as patient experience clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
Drug: Trametinib — Treatment will be administered as long as patient experience clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.

SUMMARY:
Recent preclinical studies suggest that combining MEK and MDM2 inhibition synergize to induce apoptosis in RAS/BRAF-mutant and TP53 wild-type CRC models. In vitro, in RKO cell lines (poorly differentiated colon carcinoma cell line resistant to single agent targeting MDM2 and MEK and BRAF inhibition), the MDM2 plus MEK inhibitor combination generated a synergistic increase in apoptotic index. In vivo, in mice harboring human RKO colon tumor xenografts the combination of MDM2 plus MEK inhibition elicited 93% decreases in tumor volume.

This trial is to conduct a single-center, Phase 1 dose escalation study of trametinib combined with HDM201 (a HDM2 inhibitor) in patients with advanced/metastatic RAS/RAF mutant and TP53 wt CRC.

DETAILED DESCRIPTION:
This trial is a Phase I dose escalation study aiming to evaluate the safety of a combined treatment associating HDM201 (escalating doses) with Trametinib (fixed dose). This study will utilize sequential and adaptive Bayesian design using the method of Time-to-event Continual Reassessment Method (CRM) to guide dose escalation and estimate the MTD.

ELIGIBILITY:
Inclusion Criteria:

* I1.Adult men and women ≥ 18 years at time of inform consent form signature.
* I2. Patients with histologically confirmed locally advanced or metastatic CRC bearing RAS (may be KRAS or NRAS or HRAS) or BRAF mutation, and TP53 wild type Note : TP53 wt status has to be determined by NGS sequencing of the full coding sequence using a tumor sample collected no longer than 36 months before inclusion.

Note: BRAF translocation are eligible.

* I3. Previously treated by at least one prior chemotherapy line of treatment in the advanced/metastatic setting.
* I4. Documented progressive disease and presence of at least one measurable lesion according to RECIST 1.1 based on screening tumor assessment.
* I5.Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* I6. Adequate organ function defined according to the following lab tests performed within 7 days before C1D1:

Bone marrow (without transfusion within 7 days) :Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Hemoglobin ≥ 9 g/ dL, Platelet count ≥ 100 x 109/L.

Coagulation: INR ≤ 1.5, aPTT ≤ 1.5 ULN. Note: patients receiving therapeutic anticoagulation should be on a stable dose for at least 7 days prior to C1D1.

Liver function: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤3 ULN (or ≤ 5.0 ULN in case of liver metastasis or hepatic infiltration), Serum bilirubin ≤ 1.5 ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤ 3 ULN is acceptable). Renal function:

Calculated creatinine clearance ≥ 50 mL/ min/1.73m2 or serum creatinine ≤1.5ULN. Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), formulae will be used for creatinine clearance calculation. Proteinuria ≤ +1 on dipstick or ≤ 1 g/24 hours.

* I7.Adequate cardiovascular function QTcF ≤470ms, Resting blood pressure systolic <160mmHg and diastolic<100mmHg, LVEF ≥50% as determined by transthoracic echocardiogram.
* I8.Presence of at least one biopsable lesion i.e. at least one lesion with a diameter ≥10 mm, visible by medical imaging and accessible to repeatable percutaneous or endoscopic sampling that permit core needle biopsy without unacceptable risk and suitable for retrieval of a minimum of three, but ideally four, cores using a biopsy needle of at least 16-gauge.

Note: RECIST target lesion are not to be biopsied.

-I9 Minimal wash out period required for prior treatments (delay from the last dose of the prior treatments to C1D1) : Any investigational drug > 28 days or five half-lives, whichever is longer, Major surgery >21 days, Note: If a patient underwent a major surgical procedure, he/she must have adequately recovered from the toxicity (i.e. wound healing) and/or complications from the intervention prior to starting therapy.

Radiotherapy > 28 days, Immunotherapy > 21 days, Chemotherapy > 14 days, Live vaccines > 28 days. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Growth factors targeting the myeloid lineage (e.g. GCSF, GM-CSF, M-CSF) > 14 days.

* I10 Patients able to swallow orally administered medication and do not have any clinically significant gastrointestinal abnormalities that may alter absorption of study drugs such as malabsorption syndrome or major resection of the stomach or bowels.
* I11 Fertile men must agree to use effective contraception from C1D1 until 4 months after the last dose of study drugs.
* I12 Women of child-bearing potential must have a negative serum pregnancy test within 7 days of first dose of study drugs and agree to use effective contraception from the date of negative pregnancy test to up to 4 months after the last dose of study drugs.
* I13 Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* I14 Patients must be covered by a medical insurance.

Exclusion Criteria:

* E1 Cancer disease considered curable with surgery or radiotherapy.
* E2 Prior exposure to HDM2 inhibitors and/or MEK inhibitors.
* E3 Presence of persisting AE related to anticancer treatments and Grade ≥ 2 according to CTCAE V5.0 except alopecia, neuropathy and biological values defined in inclusion criteria.
* E4 Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection that requires nutritional support).
* E5 Patients with significant active or uncontrolled cardiovascular disease or prior medical cardiac function disorders including for example uncontrolled hypertension, peripheral vascular disease, congestive heart failure (Class III-IV according to New York Heart Association [NYHA] scale), cardiac arrhythmia, or acute coronary syndrome within 6 months of C1D1 or myocardial infarction, angina pectoris, symptomatic pericarditis, within 12 months of C1D1 and patients with drug eluting stents for cardiovascular purposes.
* E6 .Patients diagnosed with treatment-related interstitial lung disease or pneumonitis.
* E7 Patients with secondary malignancy unless this malignancy is not expected to interfere with the evaluation of study endpoints and is approved by the sponsor. Examples of the latter include :basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, localized prostate cancer, prior malignancy and no evidence of disease for ≥ 2 years.
* E8 Patients requiring the use of the following forbidden concomitant treatments :

Any anticancer therapy other than the protocol specified therapies including any investigational agent, any chemotherapy, radiotherapy (except palliative radiotherapy after discussion with the sponsor), immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.

Strong and moderate inducers and inhibitors of CYP3A4/5, Live vaccines, CYP3A4/5 substrates with a narrow therapeutic index: prohibited 24 hours prior and 1 week after HDM201 administration, Substrates of OATP1B1: prohibited 24 hours prior and 48 hours after HDM201 administration.

* E9 History or current evidence of Retinal Vein Occlusion (RVO) or central serous retinopathy (CSR) or risk factors including uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes.
* E10 Patients with active hemolysis.
* E11 Known VIH infection
* E12 Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* E13 Symptomatic CNS metastases. Note: Patients with CNS metastases are eligible only if they are asymptomatic, off corticosteroids, radiographically stable for at least 2 months prior C1D1 and considered not to be at risk of bleeding.
* E14 Hypersensitivity to trametinib or HDM201 or any of their excipients.
* E15 Pregnant or breast-feeding female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Part1: Dose Maximum Tolerated | During the first 2 cycles of tratment (1 cycle = 28 days)
  A DLT is defined as occurring during the first 2 cycles of treatment and considered by the Investigator to be clinically significant and related to study drugs HDM201 and/or Trametinib, and including: Non-hematological AE as follows (Grade ≥4 non-laboratory toxicity) Grade ≥3 non-laboratory toxicity lasting > 7 days despite optimal supportive care; Any Grade ≥3 laboratory value if (Medical intervention is required to treat the patient, or, The abnormality leads to hospitalization, or The abnormality persists for > 7 days) Hematological AE as follows (Grade 4 toxicity lasting ≥ 7 days, or, Grade ≥ 3 thrombocytopenia if associated with bleeding and requires platelet transfusion, or Febrile neutropenia Grade 3 or Grade 4) Any Grade 5 related to study drugs.
  Any other study drugs related AE considered significant enough to be qualified as DLT in the opinion of the investigators after discussion with the Sponsor.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 8 weeks
  The objective response rate (ORR) after 8 weeks of treatment will be defined as the proportion of patients with complete response (CR) or partial response (PR). It will be described on the efficacy-evaluable population, together with its 95% CI. Tumor response will be evaluated according to RECIST 1.1.
Objective response rate (ORR) | 16 weeks
  The objective response rate (ORR) after 16 weeks of treatment will be defined as the proportion of patients with complete response (CR) or partial response (PR). It will be described on the efficacy-evaluable population, together with its 95% CI. Tumor response will be evaluated according to RECIST 1.1.
The duration of response (DoR) | 12 months
  The duration of response (DoR) will be measured from the time of first documented response (CR or PR as per RECIST 1.1) until the first documented disease progression or death due to underlying cancer, or censored at the date of the last available tumor assessment.
The clinical benefit rate (CBR) | 8 weeks
  after 8 weeks of treatment will be defined as the proportion of patients with CR or PR or Stable disease (SD). It will be described on the efficacy-evaluable population, together with its 95% CI. Tumor response will be evaluated according to RECIST 1.1.
The clinical benefit rate (CBR) | 16 weeks
  after 16 weeks of treatment will be defined as the proportion of patients with CR or PR or Stable disease (SD). It will be described on the efficacy-evaluable population, together with its 95% CI. Tumor response will be evaluated according to RECIST 1.1.
Progression-Free Survival (PFS) | 12 months
  will be measured from C1D1 until the date of event defined as the first documented progression or death from any cause. Patients with no event at the time of the analysis will be censored at the date of the last available tumor assessment. PFS will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CASSIER, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

IPD SHARING:
Plan to Share IPD: No